CLINICAL TRIAL: NCT07256041
Title: Play to Learn: A Comparison of Puzzle-Based and Kahoot-Based Gamification in Midwifery Education
Brief Title: Comparison of Gamification Approaches in Midwifery Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Rumeysa ÖZAYABAKAN, Asst. Prof., Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Agri Ibrahim Cecen Uni.
Record Dates: First submitted 2025-11-18; First posted 2025-12-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Education; Midwifery Education; Gameifaction
Keywords: midwifery education; gameifaction; gaming experience; puzzle; Kahoot; learning motivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puzzle Group (Experimental): A 20-question puzzle, prepared by the researchers and validated through expert opinions from 10 academic midwifery instructors using the Content Validity Index (CVI), will be distributed to the students in this group. Students will be given 10 minutes to complete the puzzle. They will solve three different puzzles at three-week intervals. Each question will be selected from the topics taught by the instructor during the preceding three weeks.
  Interventions: Other: Puzzle
- Kahoot Group (Experimental): Students in this group will form the Kahoot group. They will answer the same questions that the puzzle group solved, via the Kahoot application. Visuals will also be used in the questions at this stage. Students will respond with short answers and will be given 10 minutes for each quiz. The application will be conducted three times at three-week intervals, as with the puzzle group. Each question will be selected from the topics taught by the instructor during the preceding three weeks.
  Interventions: Other: Kahoot

INTERVENTIONS:
Other: Puzzle — Students in this group will solve three different puzzles, each administered at three-week intervals.
  Arms: Puzzle Group
Other: Kahoot — Students in this group will complete three different Kahoot quizzes, each conducted at three-week intervals.
  Arms: Kahoot Group

SUMMARY:
The aim of this study is to compare the effects of puzzle-solving and Kahoot-based learning methods on learning motivation and gaming experience among second-year midwifery students, and to evaluate students' satisfaction levels regarding these methods. The study is designed as a randomized controlled experimental research. It will be conducted between November and December 2025 with second-year students studying in the Department of Midwifery, Faculty of Health Sciences, Ağrı İbrahim Çeçen University.

The entire class will be randomly divided into two groups: Experiment 1 (Puzzle) and Experiment 2 (Kahoot). Data collection tools include the Learning Motivation Scale in Higher Education, the Gaming Experience Scale, a Satisfaction Questionnaire, Game (Kahoot-Puzzle) Achievement Test, and a Personal Information Form. For data analysis, paired-samples t-test, ANOVA, and independent-samples t-test will be used as appropriate.

DETAILED DESCRIPTION:
The lectures will be delivered by the instructor in three-week topic blocks. After each three-week block, the following procedures will be implemented:

Experiment 1 group: A 20-question puzzle prepared by the researchers and validated through expert opinions from 10 academic midwifery instructors using the Content Validity Index (CVI) will be distributed. Students will be given 10 minutes to complete the puzzle.

Experiment 2 group: The same questions will be answered via the Kahoot application.

The interventions will be conducted three times in total (e.g., during the 3rd, 6th, and 9th weeks). To prevent contamination, the groups will meet in separate classrooms, and students' phones will be collected at the entrance.

The Personal Information Form will be administered at the pre-test stage. The Learning Motivation Scale in Higher Education will also be applied as a pre-test and post-test. The Gaming Experience Scale will be administered after the first and last game sessions. The Satisfaction Scale and the Game (Kahoot-Puzzle) Achievement Test (scores obtained from the puzzle or Kahoot) will be completed after each game session.

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year midwifery student
* Enrolled in the prenatal care course
* Owning a smartphone (for the Kahoot group)
* Willingness to participate in the study
* Regular attendance in the course

Exclusion Criteria:

* Unwillingness to participate in the study
* Presence of learning disorders such as dyslexia
* Insufficient attendance in the course
* Previous participation in a similar study (Students who meet the exclusion criteria will be excluded from the study, but will continue to participate in the game activities. It is anticipated that their removal from the study could affect their performance in the course. Therefore, the scale scores of these students will not be included in the study analyses.)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | The form will be administered at the pre-test during students' first participation in the study.
  This is a 6-item form that includes questions about students' demographic characteristics, academic grade point averages, and gaming experience
Learning Motivation Scale in Higher Education (YÖMÖ-Ü) | Pre-test: Administered immediately before the first game session (on the same day). Post-test: Administered immediately after the final game session (on the same day).
  The scale consists of three sub-dimensions: learning goals, approach goals, and avoidance goals, and validity and reliability analyses have shown that it is a reliable measurement tool for Turkish university students. Each sub-dimension is scored separately, and a total score is not calculated. The scores obtained from the sub-dimensions are evaluated separately to determine which behaviors motivate students toward learning.
Gaming Experience (GAMEX) Scale | Pre-test: Administered immediately after the completion of the first game session (on the same day). Post-test: Administered immediately after the completion of the final game session (on the same day)
  The scale consists of 27 items, each scored on a 1-5 Likert scale. Items in the "Absence of Negative Effects" sub-dimension (3 items) are reverse-coded. The total score obtainable from the scale ranges from 27 to 135. Except for the "Absence of Negative Effects" sub-dimension, higher scores in the other sub-dimensions indicate a better gaming experience
Satisfaction Questionnaire | It will be completed immediately after the final game session (on the same day)
  Developed by the researchers based on the literature. Students' perceptions of the learning method will be evaluated using this questionnaire
Game (Kahoot-Puzzle) Achievement Test | Administered immediately after each game session (three time points: pre-test, mid-test, post-test) on the same day.
  Each session will include 20 prepared questions. Since the test will be scored out of 100 points, each correct answer will be worth 5 points. The scores from the games administered in the three sessions will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rumeysa ÖZAYABAKAN, Principal Investigator — Agri Ibrahim Cecen University; Betül Uncu, Principal Investigator — Istanbul University - Cerrahpasa; Rukiye DUMAN, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ağrı İbrahim Çeçen Üniversitesi, Ağrı, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided